CLINICAL TRIAL: NCT06655129
Title: Post Market Clinical Study of an Intense Pulsed Light (IPL) Medical Device as Treatment for Patient Suffering From Skin Disorder
Brief Title: Intense Pulsed Light (IPL) Medical Device as Treatment for Patient Suffering From Skin Disorder
Acronym: Anthelia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eurofeedback (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13330805
Record Dates: First submitted 2024-04-23; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Excessive Hairiness; Vascular Lesion; Pigmented Lesions; Acne Vulgaris
MeSH Terms: conditions — Hirsutism; Acne Vulgaris | interventions — Intense Pulsed Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intense Pulsed Light Treatment (Experimental): Patients will be treated at different visits, and according to the IFU, with the Anthelia Medical Device (Intense Pulsed Light).
  Interventions: Device: intense pulsed light

INTERVENTIONS:
Device: intense pulsed light — intense pulsed light (IPL) using the Medical Device Anthelia

SUMMARY:
The first IPL device obtained United States Food and Drug Administration (FDA) clearance in 1995 for treatment of lower extremity telangiectasias. Since then, its favorable cost and versatility in contrast to many singlespectrum lasers, has led to its rapid proliferation and use in a number of different clinical settings. As described in the literature, ANTHÉLIA medical device is intended to treat skin disorders:

* Excessive Hairiness (Hirsutism, Hypertrichosis...)
* Vascular lesions (Rosacea….)
* Pigmented lesions (Lentigo et melasma)
* Acne vulgaris

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women
* Excessive Hairiness:
* Patient with unwanted hair on the body (legs, arms, bikini line, or axilla)
* Patient over 18 years.
* Patients with Fitzpatrick skin types from I to V.
* Women were required to be post-menopausal, surgically sterilized, or under a medically acceptable form of birth control (i.e., oral contraceptives, IUD, contraceptive implant, or barrier methods with spermicide or abstinence) during the study time period.

Vascular lesions:

* Patients over 18 years.
* Patients with Fitzpatrick skin types from I to IV.
* Patients with varicosities and Rosacea on the face or upper and lower limbs.

Pigmented lesions:

* Patients over 18 years.
* Patients with solar lentigines on their cheeks, back, hands, arm and leg (> 3 mm).
* Patient with Fitzpatrick skin type from I to IV.

Acne:

* Patients over 18 years
* Patients with Fitzpatrick skin types from I to IV.
* Patients with facial acne vulgaris on face.
* Willing to sun protect treated area for the duration of enrollment in the study and 4 weeks after treatment.

Exclusion Criteria:

* Patients with history of malignant lesions or pre-malignant lesions, scarring, or infection in the area to be treated History of keloidal or hypertrophic scarring
* Patients with a known photosensitivity
* Pregnancy women
* Patient with diabetes mellitus suntan in the area to be treated
* Use of photo-sensitizing products for 7 days before treatment (selftanning lotions, activators, self-tanning shower gel, etc.)
* Exposure to the sun or UV rays at least 4 weeks before the treatment and 1 week afterwards
* Zones with uncovered tattoos, suspect spots or skin diseases (including spots, inflammation, beauty spots, tumors or melanomas, psoriasis, herpes...)
* Use of medication that induces anticoagulative medication or thromboembolic condition
* Patients with pacemaker or internal defibrillator
* Patients that used of NSAIDS two weeks prior to or 2 weeks following the treatment
* Epileptic patients
* Additional criteria for excessive hair: Patients that use waxing or other methods of photo epilation within 1 month prior to treatment.
* Additional criteria for acne: Patients currently under oral antibiotic or oral therapy for acne.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Efficacity for Excessive Hairiness: | up to 18 months
  Excessive Hairiness by hair counting a 4cm2 surface (To demonstrate a hair reduction of 50% between the average score of the treated aera before and after a cycle of treatment defined as six sessions spaced by 12 weeks)
Efficacity for Vascular lesions and Pigmented lesions | up to 4 months
  Vascular lesions: To demonstrate a reduction of 70% between the average score of the treated aera before and after a cycle of treatment defined as five sessions spaced by 4 weeks.
  To demonstrate a clinical improvement of 50% between the average score of the treated aera before and after a cycle of treatment defined as five sessions spaced by 4 weeks.
  Pigmented Lesions: To demonstrate a reduction of 60% between the average score of the treated aera before and after a cycle of treatment defined as three sessions spaced by 10 weeks.
Efficacity for Acne vulgaris | up to 4 months
  measuring the diameter of each pimple in a treated area (before and after), To demonstrate a lesion reduction of 50% between the average score of the treated aera before and after a cycle of treatment defined as five sessions spaced by 2 weeks.

SECONDARY OUTCOMES:
For all patients decrease of the IRBMS score | 4 to 18 months
  IRBMS (Rosenberg Self-Esteem Scale), minimum score is 10, maximum score is 40
- For all patients decrease of the DLQI score | 4 to 18 months
  DLQI (Dermatology Life Quality Index), minimum score is 0, maximum score is 30
For only Acne patients, at least 20% reduction in the ECLA score | 4 to 18 months
  ECLA ("Echelle de Cotation des Lésions d'Acné" or Acne Lesion Score Scale), minimum score is 0, maximum score is 36

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CH Auxerre, Auxerre
  - HIACT Brest, Brest
  - Centre TrialAzur, Nice
  - CH Périgueux, Périgueux
  - CHU POitiers, Poitiers

IPD SHARING:
Plan to Share IPD: No